CLINICAL TRIAL: NCT00618852
Title: A Randomized Controlled Trial of Furosemide to Prevent Fluid Overload During Red Blood Cell Transfusion in Neonates
Brief Title: Using Furosemide to Prevent Fluid Overload During Red Blood Cell Transfusion in Neonates
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Patrick McNamara/Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000009083
Record Dates: First submitted 2008-02-07; First posted 2008-02-20 (Estimated); Last update posted 2008-02-20 (Estimated); Status verified 2008-02

CONDITIONS: Lung Disease
Keywords: Pediatrics; Erythrocyte Transfusion; Furosemide; Fluid Overload
MeSH Terms: conditions — Lung Diseases; Edema | interventions — Furosemide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Furosemide
  Interventions: Drug: Furosemide
- 2 (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Furosemide — The dose of furosemide will be 1 mg/kg by intravenous bolus injection
  Arms: 1
Drug: Saline — 1 mg/kg by intravenous bolus injection
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the effects of intravenous furosemide on cardio-respiratory performance in neonates receiving a packed red blood cell (PRBC) transfusion who are considered at high risk of volume overload.

DETAILED DESCRIPTION:
Red cell transfusion is a very common practice in neonates, particularly in preterm infants. It has been estimated that approximately 300,000 neonates undergo transfusions annually. The decision to administer a blood transfusion to a sick anemic neonate is made after consideration of multiple clinical factors, including: poor weight gain, oxygenation failure, and recurrent apnea and bradycardia. These decisions are also influenced by physician preferences. For many years, furosemide has been used routinely by physicians during and after blood transfusions in neonates and other age groups. The rationale behind this common practice is to reduce the vascular overload that may be imposed by the additional blood volume delivered during transfusion. This belief, however, lacks the support of scientific clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Less than 44 weeks corrected gestational age
* Receiving a red cell transfusion
* Satisfy one of the following criteria:

  * Echocardiographic evidence of a hemodynamically significant ductus arteriosus (HSDA) defined by a transductal diameter >1.5 mm and unrestrictive systemic-pulmonary trans-ductal flow
  * Clinical evidence of significant lung disease defined by a need for respiratory support (assisted ventilation or nasal CPAP) and oxygen supplementation after 28 days of age

Exclusion Criteria:

* Infants with multiple congenital anomalies or renal insufficiency
* Infants with hypotension, hypertension, or on any cardiac medication
* Infants with sepsis causing compromised clinical condition such as disseminated intravascular coagulopathy
* Infants with contra-indications to diuretic therapy, such as significant electrolyte imbalance, or endocrine disease

Ages: 1 Week to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-12 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Cardiac chamber volume loading. | 4 hours after drug administration and 24 hours post recruitment

SECONDARY OUTCOMES:
Clinical cardio-respiratory stability (heart rate, blood pressure, respiratory rate, oxygen saturation, and oxygen requirement). | 4 hours after drug administration and 24 hours post recruitment
Myocardial performance, cardiac input and output and pulmonary hemodynamics (echocardiograph exam). | 4 hours after drug administration and 24 hours post recruitment
Changes in electrolyte balance, body weight and urine output. | 4 hours after drug administration and 24 hours post recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McNamara, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario